CLINICAL TRIAL: NCT05569967
Title: COMPARISON OF THE EFFECTS OF TELEREHABILITATION AND FACE-TO-FACE SPINAL STABILIZATION TRAININGS ON GAIT BIOMECHANICS, BALANCE AND JOINT POSITION SENSE IN TRANSTIBIAL AMPUTEES: A RANDOMIZED CONTROLLED, SINGLE BLIND STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-986/12
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Amputation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Individuals in this group will receive spinal stabilization training through telerehabilitation.
  Interventions: Other: Spinal stabilization training through telerehabilitation
- Group 2 (Active Comparator): Individuals in this group will receive spinal stabilization training face-to-face.
  Interventions: Other: Spinal stabilization training face-to-face

INTERVENTIONS:
Other: Spinal stabilization training through telerehabilitation — Individuals in both groups will receive spinal stabilization training 3 times a week for 8 weeks.
  Arms: Group 1
Other: Spinal stabilization training face-to-face — Individuals in both groups will receive spinal stabilization training 3 times a week for 8 weeks.
  Arms: Group 2

SUMMARY:
After transtibial amputations, biomechanical changes in the trunk, pelvis, and lumbar region cause asymmetrical strength and core muscle activation on the amputated side, which negatively affects the gait biomechanics of individuals. However, routine treatment programs do not use treatment approaches based on the core region. This study will focus on the effects of telerehabilitation and face-to-face spinal stabilization exercise training on gait, balance, joint position sense, core muscle function, and perceived mobility in transtibial amputees, after treatment, and after long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who use total contact sockets
* have been using prostheses for at least 1 year,
* can walk independently without a walking aid
* functionally at least K2

Exclusion Criteria:

* Bilateral amputation
* Upper extremity amputation
* Neurological problems
* Other orthopedic problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
gait speed | Change from baseline at 8 weeks and 5 months
  Participants will be asked to walk on flat ground for 10 meters. At this time, the speed will be evaluated by the BTS G-Walk sensor.

SECONDARY OUTCOMES:
spatial parameter of gait | Change from baseline at 8 weeks and 5 months
  Participants will be asked to walk on flat ground for 10 meters. At this time, the spatial variable of gait will be evaluated by the BTS G-Walk sensor.
temporal parameter of gait | Change from baseline at 8 weeks and 5 months
  Participants will be asked to walk on flat ground for 10 meters. At this time, the temporal variable of gait will be evaluated by the BTS G-Walk sensor.
Dynamic Balance | Change from baseline at 8 weeks and 5 months
  Dynamic balance; will be evaluated with the "Four Square Step Test", which is a valid and reliable measure in the evaluation of gait, mobility and dynamic balance. The time to complete four frames is recorded. If the duration is more than 24 seconds, it is considered that there is a risk of falling.
Balance confidence | Change from baseline at 8 weeks and 5 months
  Balance confidence of individuals will be evaluated with the "Activity-Specific Balance Confidence Scale". On this scale, individuals score their balance confidence between 0% and 100% during various ambulatory activities. A mean score of 50% or less indicates low physical function, 50-80% indicates moderate physical function, and 80% or higher indicates high physical function.
Core Muscle Strength | Change from baseline at 8 weeks and 5 months
  The strength of the core muscles will be evaluated using "The Stabilizer Pressure Biofeedback Unit". The pressure values for the measurement will be recorded 3 times in a row, at the beginning and end of the 10-second contraction, and the average value will be taken.
Core Muscle Endurance- Trunk Flexor | Change from baseline at 8 weeks and 5 months
  The trunk flexor test will be performed with the arms crossed over the thorax, the trunk at 55 degrees of flexion, and the knees and hips flexed to 90 degrees. The test will be finished when the participant is unable to maintain the position. The time will be recorded.
Core Muscle Endurance- Trunk Extansor | Change from baseline at 8 weeks and 5 months
  The trunk extensor test will be performed in the prone position, with the pelvis, hips and knees fixed to the bed. The participant will be asked to cross his arms over his body and position his body horizontally. The test will be finished when the participant is unable to maintain the horizontal position. The time will be recorded.
Core Muscle Endurance- Side Bridge | Change from baseline at 8 weeks and 5 months
  While the participants are in the side-lying position, they will raise their hips and align their bodies in a straight line by getting support from their feet and elbows. The time will be recorded by asking them to maintain the position as much as possible.
Perceived Mobility | Change from baseline at 8 weeks and 5 months
  The Prosthetic Limb Users Survey of Mobility (PLUS-M) Short Form will be used. The questionnaire consists of a total of 12 items, each of which is evaluated over 0-5 points. All items evaluate the degree of ability of the individual to perform the activity rather than the actual performance of the individual, and reflect the difficulty experienced by the individual while performing the activity. Higher scores indicate better mobility.
Joint Position Sense-Knee | Change from baseline at 8 weeks and 5 months
  It will be evaluated with a dual digital inclinometer (ACUMAR™).While the participants are in the prone position, the inclinometer will be placed on the femur and fibula and they will be asked to flex the knee at 40 degrees. It will be asked to feel the angle completely by keeping it in this position for a certain period of time and then return to the neutral position. The patient will then be asked to find the target angle. The difference between the target angle and the obtained angle will be determined as an absolute value and recorded in degrees.
Joint Position Sense-Trunk | Change from baseline at 8 weeks and 5 months
  It will be evaluated with a dual digital inclinometer (ACUMAR™). The test will be performed in a standing position with eyes closed, barefoot on a hard floor, with the support surface shoulder-width apart. The inclinometer will be fixed on the T1 and S1 spinous processes and 30 degrees of trunk flexion will be required. It will be asked to feel the angle completely by keeping it in this position for a certain period of time and then return to the neutral position. The patient will then be asked to find the target angle. The difference between the target angle and the obtained angle will be determined as an absolute value and recorded in degrees.
pelvic parameter of gait | Change from baseline at 8 weeks and 5 months
  Participants will be asked to walk on flat ground for 10 meters. At this time, the pelvic parameter of gait will be evaluated by the BTS G-Walk sensor.
Step symmetry | Change from baseline at 8 weeks and 5 months
  The time-distance characteristics of the gait will be used to calculate the gait symmetry. The step time of the non-amputee will be calculated in proportion to the amputated side.
Stance symmetry | Change from baseline at 8 weeks and 5 months
  The time-distance characteristics of the gait will be used to calculate the gait symmetry. The stance time of the non-amputee will be calculated in proportion to the amputated side.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)